CLINICAL TRIAL: NCT07207408
Title: Phase 2, Randomized, Multicenter Trial of the Immunogenicity, Safety, and Tolerability of rF1V-1018 Vaccine in Adults 18 to 55 Years of Age
Brief Title: Immunogenicity, Safety, and Tolerability of rF1V-1018 Vaccine in Adults 18 to 55 Years of Age
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DV2-DC02-02
Record Dates: First submitted 2025-10-02; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Prevention of Pneumonic Plague Resulting From Aerosol Exposure to Yersenia Pestis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is partially blinded which means observers and participants know what study vaccine is being administered for some treatment arms but not for other treatment arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Experimental)
  Interventions: Biological: rF1V-1018
- Arm 2 (Experimental)
  Interventions: Biological: rF1V-1018
- Arm 3 (Experimental)
  Interventions: Biological: rF1V-1018
- Arm 4 (Experimental)
  Interventions: Biological: rF1V-1018
- Arm 5 (Experimental)
  Interventions: Biological: rF1V-1018
- Arm 6 (Experimental)
  Interventions: Biological: rF1V-1018

INTERVENTIONS:
Biological: rF1V-1018 — Regimen 1
  Arms: Arm 1
Biological: rF1V-1018 — Regimen 2
  Arms: Arm 2
Biological: rF1V-1018 — Regimen 3
  Arms: Arm 3
Biological: rF1V-1018 — Regimen 4
  Arms: Arm 4
Biological: rF1V-1018 — Regimen 5
  Arms: Arm 5
Biological: rF1V-1018 — Regimen 6
  Arms: Arm 6

SUMMARY:
This study will evaluate the immunogenicity, safety, and tolerability of rF1V-1018 vaccine

DETAILED DESCRIPTION:
This dose-finding study will evaluate the immunogenicity, safety, and tolerability of multiple doses and regimens of rF1V-1018 vaccine in healthy adults. Immunogenicity blood samples will be drawn at several timepoints during the study. Participants will return to the clinic for periodic visits for study specific evaluations including evaluation of immunogenicity and safety. Safety assessments will be done at regular intervals through the end of the trial.

Six dose regimens will be tested in Part 1 of the study. Up to two dose regimens from Part 1 will be chosen for Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 55 years of age
2. Healthy participants or participants with stable pre-existing medical conditions Pre-existing stable medical condition means a participant who: has full capacity of daily activity and no major medication modification within 3 months prior to Day 1; has not undergone surgical or minimally-invasive intervention or had any hospitalization/emergency room visit for the specific medical condition.
3. Able to comply with the protocol schedule and procedures
4. Able and willing to provide written informed consent
5. If female of child-bearing potential and heterosexually active, has practiced adequate contraception for at least 28 days prior to vaccination, has negative pregnancy tests just prior to vaccination, and has agreed to continue adequate contraception through three months following the final trial injection

A premenopausal woman who has at least one of the following is considered not of childbearing potential:

1. Documented hysterectomy
2. Documented bilateral salpingectomy
3. Documented bilateral oophorectomy
4. Documented and current bilateral tubal ligation or occlusion

Exclusion Criteria:

1. A history of plague disease or have previously received any plague vaccine
2. Active tuberculosis or other systemic infectious process
3. History of human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV) infection, or positive test for antibody to HIV, HBV, or HCV
4. History of autoimmune disorder
5. History of sensitivity to any component of trial vaccines
6. Body mass index ≥ 30 kg/m2
7. Has received the following prior to any trial injection:

   a) ≤ 14 days: i) Any licensed or authorized inactivated vaccines (including vaccines containing mRNA or CpG) b) ≤ 28 days: i) Any live vaccine ii) Any investigational medicinal agent c) ≤ 90 days: i) Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the first trial vaccine administration or planned administration during the trial period. (For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent). Inhaled, topical, and intraarticular steroids are allowed.

   ii) Granulocyte or granulocyte-macrophage colony stimulating factor iii) Immunoglobulins or any blood products (receipt of certain monoclonal antibodies may on a case-by-case basis be non-exclusionary if approved via consultation with Sponsor Medical Monitor) iv) Antisense oligonucleotides v) Drugs/investigational agents with very long half-lives (defined as ≥ 60 days) (eg, radioactive iodine, amiodarone, liraglutide, nirsevimab, teplizumab, evinacumab, and obinutuzumab) vi) Infusion of blood products d) At any time: DNA plasmids or other genetic therapy intended to integrate permanently into host cells
8. If female is pregnant (known before or established at the time of screening), breastfeeding, or planning breastfeeding or a pregnancy
9. Is undergoing chemotherapy or expected to receive chemotherapy during the trial period; has a diagnosis of cancer within the last 5 years other than squamous cell or basal cell carcinoma of the skin
10. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
11. Oral temperature ≥ 38°C (≥ 100.4°F) at the time of vaccine administration
12. History of acute myocardial infarction (AMI) or documented coronary artery disease (CAD)

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Anti-rF1V antibody level | 4 weeks after final study vaccine
Evaluate safety of rF1V-1018 | injection reactions through 7 days after each study vaccine, adverse events for 28 days after each study vaccine; SAEs, MAEs, imAESIs through 6 months after the final study vaccine
  Evaluate adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - AMR- Miami, Miami, Florida
  - AMR- El Dorado, El Dorado, Kansas
  - AMR- Las Vegas, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No